CLINICAL TRIAL: NCT06039527
Title: TINO: Identifying the Underlying Mechanisms and Consequences of the Loss of Nasal T Cells in Vital and Frail Older Individuals
Brief Title: TINO: T Cells in the Nose of Older Adults
Acronym: TINO
Status: Recruiting | Type: Observational
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, Simon P Jochems, PhD, Assistant professor, Leiden University Medical Center
Other Study IDs: P21.066; NL77841.058.21 (Registry Identifier: toetsingonline.nl)
Record Dates: First submitted 2023-09-01; First posted 2023-09-15 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Respiratory Tract Infections; Aging
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Investigators will collect the following samples:
  * peripheral blood
  * nasopharyngeal swab
  * oropharyngeal swab
  * nasal curettes
  * nasosorption
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Young adults: N=50 of this group No intervention. Sampling at timepoint 0 and for 50% of the group another sample at 3 months If respiratory symptoms develop in the 3 months after timepoint 0, participants are invited to provide a NPS/OPS to identify causative agent, and if one is established, individuals are sampled 3 more times at months 1, 3 and 5 post symptom onset
- Vital elderly: N=60 of this group No intervention. Sampling at timepoint 0 and for 50% of the group another sample at 3 months If respiratory symptoms develop in the 3 months after timepoint 0, participants are invited to provide a NPS/OPS to identify causative agent, and if one is established, individuals are sampled 3 more times at months 1, 3 and 5 post symptom onset
- Frail elderly: N=60 of this group. Half with recurring respiratory infections, and half without No intervention. Sampling at timepoint 0 and for 50% of the group another sample at 3 months If respiratory symptoms develop in the 3 months after timepoint 0, participants are invited to provide a NPS/OPS to identify causative agent, and if one is established, individuals are sampled 3 more times at months 1, 3 and 5 post symptom onset

SUMMARY:
Rationale: Individuals with advanced age are at a progressively increasing risk of acquiring lower respiratory tract infections. Besides calendar age, the degree of frailty also associates with increased susceptibility to pneumonia requiring hospitalization. How alterations in the mucosal immune system with advanced age predispose to infections remains unclear as access to relevant tissue samples is limited. With minimally-invasive nasal sampling methods, it was recently observed that in vital older adults, both CD4+ T cells and CD8+ T cells are selectively lost from the nasal mucosa. However, the exact phenotype, underlying mechanisms, key molecules and consequences of this have not yet been investigated.

Objective:

Elucidate the mechanisms underlying the loss of nasal T cells and characterize in depth the differences of T cells in young and older adults and associate this loss with susceptibility to infections.

Study design: Prospective cohort study

Study population: Participants will be recruited from 3 groups:

* healthy young adults (18-30 years, n=50)
* vital older adults (>65 years, n=60)
* frail elderly (>65 years, n=60). This group includes individuals without a history of recurrent respiratory infections or with >2 self-reported episodes of respiratory infection in the past year.

Main study parameters/endpoints: Frequency of nasal CD8+ T cells in young adults and frail older adults.

Secondary study parameters/endpoints:

* Phenotype (subsets, activation status), functionality, transcriptomic state, clonality and frequency of nasal and blood T cell populations
* Stability of T cells and other immune parameters, as described for main study parameter, during a second sample after 3 months.
* Analysis of other immune populations as for main study parameter
* Concentration of nasal and systemic factors (e.g. cytokines and metabolites) and their association with T cells and other immune populations
* Respiratory tract microbiota profiles and presence of asymptomatic viral infections and their association with T cells and other immune parameters
* Chronological and biological age, sex, and other immunologically relevant parameters with T cell populations and other immune parameters
* Alteration of T cell phenotype, during and following respiratory tract infections. Levels of antigen-specific T cells and other immune parameters in nose and blood post infection.

ELIGIBILITY:
Inclusion Criteria:

•Adults able and willing to provide informed consent.

Specific inclusion criteria per group:

* Young adults aged 18-30 years old
* Healthy elderly aged >65 years old
* Frail elderly >65 years old
* Clinical Frailty score healthy elderly 1-3
* Clinical Frailty score frail elderly >3
* Self-reported respiratory tract infection in previous year healthy elderly 0-1
* Self-reported respiratory tract infection in previous year frail elderly 0-1 or >1

Exclusion Criteria:

* Incompetence to provide informed consent prior or during study
* Current smoker or >40 pack year history
* History of severe nose bleedings
* Diagnosed with asthma, COPD or chronic rhinosinusitis
* Use of inhalation corticosteroids or antibiotics in the past 6 weeks
* Current use of anti-coagulants (to prevent nosebleeds). Platelet inhibitors like acetylsalicylzuur (Ascal) are allowed.
* Respiratory tract infection or common cold in the past 2 weeks
* Immunocompromised individuals (with primary immune deficiency or secondary immune deficiency)
* Life expectancy <28 days in the opinion of study physician
* Vaccination in the 2 months prior to study start. A potential subject that is only excluded from participation based on a recent vaccination will be asked to re-participate 2 months post vaccination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study population: Investigators will recruit participants from 3 groups:
  * healthy young adults (18-30 years, n=50)
  * vital older adults (>65 years, n=60)
  * frail elderly (>65 years, n=60). These will be consist of individuals without a history of recurrent respiratory infections or with >2 self-reported episodes of respiratory infection in the past year.
  Frailty will be determined by a clinical frailty score. The Clinical Frailty Scale (CFS) is a scale that caretakers can use to identify level of frailty in older patients from 1 (very fit) through 9 (terminally ill). For the present study, "vital older patients" are defined as those with a CFS of 1-3 and "older patients living with frailty with a CFS of 4 or higher".
Sampling Method: Non-Probability Sample
Enrollment: 170 (Estimated)
Dates: Start 2021-01-24 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Frequency of nasal CD8+ T cells in young adults and frail older adults. | baseline sample or month 3 sample
  CD8 T cells relative to nasal epithelial cells (ratio)

SECONDARY OUTCOMES:
Phenotype of nasal and blood T cell populations in young adults, healthy older adults and frail older adults that suffer from recurrent respiratory tract infections or not. | baseline sample or month 3 sample
  percentage of T cells and T cell subsets
Functionality of nasal and blood T cell populations in young adults, healthy older adults and frail older adults that suffer from recurrent respiratory tract infections or not. | baseline sample or month 3 sample
  percentage of T cells responding to in vitro stimulations
Transcriptomic cluster composition of nasal and blood T cell populations in young adults, healthy older adults and frail older adults that suffer from recurrent respiratory tract infections or not, as frequency of T cell subsets. | baseline sample or month 3 sample
  T cell clusters based on gene expression patterns
Clonality of nasal and blood T cell populations in young adults, healthy older adults and frail older adults that suffer from recurrent respiratory tract infections or not. | baseline sample or month 3 sample
  Number and proportion of TCR clones
Stability of nasal T cells, as described for main study parameter, during a second sample after 3 months. | baseline sample versus month 3 sample
  CD8 T cells relative to nasal epithelial cells (ratio)
Stability of nasal immune populations, during a second sample after 3 months. | baseline sample versus month 3 sample
  immune cell populations relative to nasal epithelial cells (ratio)
Comparison of nasal immune cell populations between young adults, vital and frail elderly | baseline sample or month 3 sample
  ratio to epithelial cells
Comparison of peripheral immune cell populations between young adults, vital and frail elderly | baseline sample or month 3 sample
  percentage of total CD45+ cells
Concentration of nasal and systemic cytokines | baseline sample or month 3 sample
  concentrations
Concentration of nasal and systemic metabolitesother immune populations | baseline sample or month 3 sample
  concentrations
Respiratory tract microbiota profiles and their association with T cells and other immune parameters | baseline sample or month 3 sample
  microbiota abundance (total sum scaling)
Presence of asymptomatic viral infections and their association with T cells and other immune parameters | baseline sample or month 3 sample
  viral of loads (Ct)
Effect of sex on aging effects of nasal immune populations | baseline sample or month 3 sample
  ratio to nasal epithelial cells
Effect of sex on aging effects of blood immune populations | baseline sample or month 3 sample
  percentage of CD45+ cells
Frequencies of antigen-specific T cells in nose post infection. | symptom onset and 1, 3 and 5 months later
  antigen-specific T cells as percentage of T cells
Frequencies of antigen-specific T cells in blood post infection. | symptom onset and 1, 3 and 5 months later
  antigen-specific T cells as percentage of T cells

CONTACTS AND LOCATIONS:
Overall Officials: Simon P Jochems, PhD, Principal Investigator — LUMC
Locations (1):
- Leiden University Medical Center, Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No
As even pseudonymized data is considered personal data as these can sometimes be traced back to an individual, data can be requested from the PI. If requests fall within the scope of the informed consent and study protocol, an MTA/DTA can be shared. Data will be posted on repositories with restricted access.